CLINICAL TRIAL: NCT01658410
Title: Short-term Endothelin A Receptor Blockade in Patients With On-pump Coronary Artery Bypass Grafting
Brief Title: Short-term Endothelin A Receptor Blockade in Patients With On-pump CABG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alfred A Kocher, MD, Professor, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-023552-90
Record Dates: First submitted 2012-07-26; First posted 2012-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease; Aorto-coronary Bypass Grafting
Keywords: Coronary artery disease; bypass grafting
MeSH Terms: conditions — Coronary Artery Disease | interventions — cyclo(Trp-Asp-Pro-Val-Leu)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BQ-123 (Active Comparator)
  Interventions: Drug: BQ-123
- NaCl (Placebo Comparator)
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: BQ-123 — BQ-123 (Clinalfa, Läufelfingen, Switzerland) Dosage: 15µmol in two equal amounts (7.5µmol); in the first and last cardioplegia Route: intracoronary
  Other Names: Cyclo(-D-Trp-D-Asp-Pro-D-Val-Leu) sodium salt
  Arms: BQ-123
Drug: NaCl — NaCl, Route: intracoronary
  Arms: NaCl

SUMMARY:
Background: Although selected cardiac surgery can be performed off-pump, the vast majority of cardiac surgical procedures today are performed with the support of cardiopulmonary bypass (CPB). Blood cardioplegia is used to protect the heart during aortic cross-clamping. However, negative effects of myocardial hypoxia during surgery are often aggravated by ischemia/reperfusion injury. In addition, cardiopulmonary bypass leads to an inflammatory response including endothelial cell activation.

Comparable to the reperfusion injury following acute myocardial infarction resolved by percutaneous coronary intervention, the microcirculatory impairment observed after cardiac surgery may be caused by endothelin 1 (ET-1). ET-1 is a potent vasoconstrictor peptide upregulated in myocardial ischemia-reperfusion injury. Short-term administration of the selective ETA receptor blocker BQ-123 was found safe in a pilot study including patients with acute myocardial infarction.

Hypothesis: Acute local ETA receptor blockade by intracoronary administered BQ-123 reduces myocardial injury.

Methods: BQ-123 will be administered in patients undergoing on-pump aorto-coronary bypass grafting to the left anterior descending coronary artery with the use a left inner mammary artery graft and at least one vein graft. Subjects will be randomized to receive the endothelin-A receptor blocker BQ-123 or placebo administered intracoronarily in combination with cardioplegia in a double-blind manner. The primary endpoint will be enzymatic infarct size.

Clinical perspective: The implementation of BQ-123 as an add-on pharmacologic therapy in cardiac surgery performed with the use of cardiopulmonary bypass could lead to improved tissue reperfusion and reduced ischemia/reperfusion injury, potentially impacting clinical long-term outcome.

DETAILED DESCRIPTION:
Background: Although selected cardiac surgery can be performed off-pump, the vast majority of cardiac surgical procedures today are performed with the support of cardiopulmonary bypass (CPB). Blood cardioplegia is used to protect the heart during aortic cross-clamping. However, negative effects of myocardial hypoxia during surgery are often aggravated by ischemia/reperfusion injury. In addition, cardiopulmonary bypass leads to an inflammatory response including endothelial cell activation.

Comparable to the reperfusion injury following acute myocardial infarction resolved by percutaneous coronary intervention, the microcirculatory impairment observed after cardiac surgery may be caused by endothelin 1 (ET-1). ET-1 is a potent vasoconstrictor peptide upregulated in myocardial ischemia-reperfusion injury. Short-term administration of the selective ETA receptor blocker BQ-123 was found safe in a pilot study including patients with acute myocardial infarction. Patients with posterior-wall STE-ACS (n=57) were randomly assigned to receive intravenous BQ-123 at 400nmol/minute or placebo over 60 minutes, starting immediately prior to primary percutaneous coronary intervention (PCI). No side branch occlusions, bleeding complications or severe systemic hypotensive episodes occurred and all patients were alive at 30 days.

Hypothesis: Acute local ETA receptor blockade by intracoronary administered BQ-123 reduces myocardial injury.

Methods: BQ-123 will be administered in patients undergoing on-pump aorto-coronary bypass grafting to the left anterior descending coronary artery with the use a left inner mammary artery graft and at least one vein graft. After a 1:1 randomized pilot safety-phase with 30 patients administering half the dose, 90 subjects will be randomized to receive 15µmol BQ-123 dissolved in NaCl 0.9% or placebo (NaCl 0.9% ) administered intracoronarily in combination with cardioplegia in a double-blind manner. The primary endpoint will be enzymatic infarct size assessed by the area under the curve of myocard specific creatine kinase-MB isoform (CK-MB). Left ventricular ejection fraction, diastolic dysfunction and, perioperative echocardiography, postoperative levels of myeloperoxidase and matrixmetalloproteinase-9 activity as well as MACE will serve as secondary endpoints.

Clinical perspective: The implementation of BQ-123 as an add-on pharmacologic therapy in cardiac surgery performed with the use of cardiopulmonary bypass could lead to improved tissue reperfusion and reduced ischemia/reperfusion injury, potentially impacting clinical long-term outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing on-pump coronary artery bypass grafting using the left mammary artery to the left anterior descendent artery and at least one vein graft due to coronary artery disease, aged 18 years and above.

Exclusion Criteria:

* Significant liver disease (Transaminases and/or gamma-GT > 3 fold upper limit)
* Glomerular filtration rate <40mL/h
* History of severe congestive heart failure (Left ventricular ejection fraction <35%)
* Current atrial fibrillation
* Significant valvular heart disease requiring valve replacement Department of Cardiac Surgery
* Primary myocardial disease
* Acute coronary syndrome or cardiogenic shock (sRR <90mmHg or need for inotropic support)
* Women with child-bearing potential
* Subjects with contraindications for CMR (cardiac magnetic resonance)
* Inability to read, understand and sign the informed consent
* Life expectancy <1y
* Prior organ transplantation
* Participation in a clinical trial using an investigational medical product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
enzymatic infarct size | 72h

SECONDARY OUTCOMES:
Catecholamines | 5h
Liver function | 72h
catecholamine requirement | 72h

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Kocher, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria, Austria